CLINICAL TRIAL: NCT00846976
Title: A Treatment Protocol to Monitor the Safety of a 200 mg Daily Dose of Bicalutamide (Casodex) in Patients With Advanced Prostate Cancer
Brief Title: Treatment Protocol to Monitor the Safety of a 200 mg Dose of Bicalutamide in Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6874C00014
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
Keywords: Safety
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 200 mg Casodex (Experimental)
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Bicalutamide — 200mg daily
  Other Names: Casodex

SUMMARY:
This is an open label, single-centered treatment protocol designed to monitor the safety of patients treated with a 200 mg daily dose of CASODEX. Patient will receive CASODEX as long as physician feels that he is benefiting from this form of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate gland
* Patients with advanced prostate cancer
* Adult male over the age of 18 years old
* Normal liver function (AST < 2 x Upper Limit Normal)

Exclusion Criteria:

* ECOG performance status of 4.
* Previous history or presence of another malignancy other than prostate cancer or treated squamous/basal cell carcinoma of the skin, within the last 5 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 1994-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety profile of patients treated with a 200 mg daily dose of CASODEX | every three months

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, New York, New York, United States

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=578&filename=CSR-D6874C00014.pdf
- See also: CSR-D6874C00014.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=578&filename=CSR-D6874C00014.pdf